CLINICAL TRIAL: NCT04433702
Title: A Controlled, Open-Label, Randomized Study to Evaluate the Application of Negative Pressure to the Periocular Microenvironment to Alter Pattern Electroretinography Readings by Way of Modulating Intraocular Pressure
Brief Title: Effect of Negative Pressure on Pattern Electroretinography Readings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed the study design and opened a new study
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CP-014
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma; Open Angle, Low Risk; Ocular Hypertension; Glaucoma Suspect
Keywords: glaucoma treatment; multi-pressure dial; pattern electroretinography; open-angle glaucoma
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental Eye (Experimental): 10 mmHg of negative pressure is applied to the periocular microenvironment. This is achieved by programming the Mercury™ Multi-Pressure Dial (MPD) such that only one goggle receives negative pressure.
  Interventions: Device: Mercury™ Multi-Pressure Dial (MPD) Experimental Goggle
- Control Eye (Placebo Comparator): The opposing eye serves as the intrasubject control for each participant. No negative pressure is applied to the periocular microenvironment. This is achieved by programming the Mercury™ Multi-Pressure Dial (MPD) such that the other goggle does not receive negative pressure.
  Interventions: Device: Mercury™ Multi-Pressure Dial (MPD) Placebo Goggle

INTERVENTIONS:
Device: Mercury™ Multi-Pressure Dial (MPD) Experimental Goggle — The Mercury™ MPD applies negative pressure to one of the two goggles inducing an IOP reduction of 10 mmHg. This is randomized for each subject in the trial.
  The Mercury™ MPD consists of:
  1. Goggles: seal against the bony orbit with straps around head. The goggles separately enclose each eye, with each eye individually connected to a pressure-modulating pump.
  2. Programmable pump: applies negative pressure inside the goggles via clear tubing attached to a handheld device
  Arms: Experimental Eye
Device: Mercury™ Multi-Pressure Dial (MPD) Placebo Goggle — The Mercury™ MPD applies no negative pressure to one of the two goggles eliciting no IOP reduction. This is randomized for each subject in the trial.
  The Mercury™ MPD consists of:
  1. Goggles: seal against the bony orbit with straps around head. The goggles separately enclose each eye, with each eye individually connected to a pressure-modulating pump.
  2. Programmable pump: applies negative pressure inside the goggles via clear tubing attached to a handheld device
  Arms: Control Eye

SUMMARY:
Glaucoma is a leading cause of blindness worldwide. Intraocular pressure (IOP) remains the only modifiable risk factor for glaucoma. Without sufficient IOP lowering therapy, glaucoma induces retinal ganglion cell death and visual field loss. Pattern electroretinography (pERG) measurements directly correlate with retinal ganglion cell (RGC) signaling, providing an objective, repeatable, and non-invasive assessment of RGC function. The purpose of the study is to investigate the pERG changes associated with acute IOP reduction using the Mercury™ Multi-Pressure Dial (MPD). 10 patients will be enrolled. These subjects will have a best corrected visual acuity of 20/40 or better in both eyes and an established diagnosis of one of either mild/moderate OAG (open-angle glaucoma), OHT (ocular hypertension), or glaucoma suspect. Both eyes will be enrolled in the study. The study eye will receive a standardized 10 mmHg decrease in periorbital pressure via the Mercury™ Multi-Pressure Dial (MPD), and the fellow/control eye will receive no (zero) pressure application. Total google wear time will be 4.5 hours. Serial pERG measurements will be taken before, immediately after, and 2 hours after negative pressure application.

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of committing to the duration of the study and signing the informed consent.
* Subjects must be male or female and ≥ 22 years of age at the time of signing the informed consent.
* Subjects with orbital anatomy that permits a proper seal when goggles are placed over eyes.
* Subjects can tolerate ERG measurements.
* Subjects with a documented BCVA OU 20/40 or better AND a diagnosis of OHT, glaucoma suspect, or OAG in both eyes. OAG definition is inclusive of normal tension glaucoma, pseudoexfoliation glaucoma, and pigment dispersion. Both eyes require same diagnosis.
* Subjects with prior surgeries such as refractive surgeries (e.g., LASIK, PRK, SMILE), cataract surgery, cataract surgery with minimally invasive glaucoma surgery (MIGS), MIGS alone, trabeculectomy, or implantation of other glaucoma drainage devices can be included in the study; however, no other prior ocular surgeries are permitted.
* Subjects without lenticular opacities and/or trace (i.e. 1+) lenticular opacities.

Exclusion Criteria:

* Subjects with a history of allergy to primary study device material (i.e. silicone, anti-fog solution).
* Subjects with a history of any ocular disorder or condition in either eye that would likely interfere with the interpretation of the study results or subject safety (e.g., corneal transplant).
* Subjects with a history of any demyelinating disorder or condition that would likely interfere with the interpretation of the study results or subject safety (e.g. MS).
* Subjects with an untreated retinal detachment, retinal tears, macular degeneration, or any other fundus findings that may prevent accurate ERG measurements in either eye.
* Subjects with conjunctival chemosis in either eye.
* Subjects with eyelid edema.
* Subjects with a history of seizure disorder.
* Subjects with an eye infection.
* Subjects with moderate-severe (i.e. 2+, 3+, or 4+) lenticular opacities.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pattern Electroretinography (pERG) Alterations | 0 hours; 4.5 hours; 6.5 hours
  Mercury™ MPD alters IOP in study eyes of subjects per controlled reduction of pressure. pERG changes induced by the Mercury™ MPD will provide insight into changes in retinal ganglion cells after wearing Mercury™ MPD with negative pressure applied anterior to the orbital rim.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Greenwood, MD, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No